CLINICAL TRIAL: NCT01626495
Title: CHP 959 - A Phase I/IIA Study of Redirected Autologous T Cells Engineered to Contain Anti-CD19 Attached to TCRzeta and 4-1BB Signaling Domains in Patients With Chemotherapy Resistant Or Refractory CD19+ Leukemia and Lymphoma
Brief Title: Phase I/IIA Study of CART19 Cells for Patients With Chemotherapy Resistant or Refractory CD19+ Leukemia and Lymphoma
Acronym: Pedi CART19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-007706, 815870; CHP959 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2012-06-18; First posted 2012-06-22 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: B Cell Leukemia; B Cell Lymphoma
Keywords: Biological: CART19
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CART-19 T Cells (Experimental): The subject's thawed T cells will be modified in one or two different ways that will allow the cells to identify and kill the tumor cells (B cells). The T cells will be infused over 10-15 minutes on days Days 0, and 1. Day 14 is tentative based on response.
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — Day 0: 10% of total dose Day 1: 30% of total dose if patient is stable (no significant toxicity) from prior dose.

SUMMARY:
This is a study for children who have been previously treated for Leukemia/Lymphoma. In particular, it is a study for people who have a type of Leukemia/Lymphoma that involves B cells (a type of white cell), which contain the cancer. This is a new approach for treatment of Leukemia/Lymphoma that involves B cells (tumor cells). This study will take the subject's white blood cells (T cells) and modify them in order to target the cancer.

The subject's T cells will be modified in one or two different ways that will allow the cells to identify and kill the tumor cells (B cells). Both ways of modifying the cells tells the T cells to go to the B cells (tumor cells) and turn "on" and potentially kill the B cells (tumor cells). The modification is a genetic change to the T cells, or gene transfer, in order to allow the modified T cells to recognize your tumor cells but not other normal cells in the subject's body. These modified cells are called chimeric antigen receptor 19 (CART19) T-cells.

DETAILED DESCRIPTION:
At entry subjects will be staged and the suitability of their T cells for CART-19 manufacturing will be determined. Subjects who have adequate T cells will be leukapheresed to obtain large numbers of peripheral blood mononuclear cells (PBMC) for CART-19 manufacturing. The T cells will be purified from the PBMC, transduced with CART-19 lentiviral vector, expanded in vitro and then frozen for future administration. Chemotherapy will then be given. Following tumor burden reassessment, CART-19 cells will be thawed and infused.

Subjects will have blood tests to assess safety, and engraftment and persistence of the CART-19 cells at regular intervals through four weeks after their last infusion of the study. Following the 6 months of intensive follow-up, subjects will be evaluated quarterly for two years with a medical history, a physical examination, and blood tests. Following this evaluation, subjects will enter a roll-over study for annual follow-up by phone and questionnaire for an additional thirteen years to assess for the diagnosis of long-term health problems, such as development of new malignancy.

Primary objectives:

1. Determine the safety and feasibility of administration of chimeric antigen receptor T cells transduced with the anti-CD 19 lentiviral vector (referred to as "CART-19" cells).
2. Determine duration of in vivio survival of CART-19 cells. Real Time polymerase chain receptor (RT-PCR) analysis of whole blood will be used to detect and quantify survival of CART-19 TCR:4-1BB and TCR cells over time.

Secondary objectives:

1. For patients with detectable disease, measure anti-tumor response due to CART-19 cell infusions.
2. To determine if the 4-1BB transgene is superior to the TCR only transgene as measured by the relative engraftment levels of CART-19 TCR:4-1BB and TCR cells over time.
3. For patients with stored or accessible tumor cells (such as patients with active chronic lymphocytic leukemia (CLL), acute lymphoblastic leukema (ALL), etc) determine tumor cell killing by CART-19 cells in vitro.
4. Determine if cellular or humoral host immunity develops against the murine anti-CD19, and assess correlation with loss of detectable CART-19 (loss of engraftment).
5. Determine the relative subsets of CART-19 T cells (Tcm, Tem, and Treg)

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with CD 19+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to <2 year survival) with currently available therapies will be enrolled:

1. Eligible diseases: CD 19+ leukemia or lymphoma

   1. ALL without curative options for therapy, including those not eligible for allogeneic

      SCT because of:
      * age
      * co-morbid disease
      * other contraindications to TBI-based conditioning (required for ALL SCT)
      * lack of suitable donor
      * prior SCT
      * Declines allo SCT (in CR3) as a therapeutic option after documented discussion about the role of SCT with a BMT physician not part of the study team. Note: Patient may be in any complete response, or patient may have active disease but responding or stable after most recent therapy. The intent is not to enroll patients with no degree of disease control, or rapidly increasing disease burden between enrollment and cell infusion.
   2. Follicular lymphoma, previously identified as CD19+

      * At least 2 prior combination chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy.
      * Stage III-IV disease.
      * Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval <1 year).
      * Disease responding or stable after most recent therapy (chemotherapy, MoAb).
   3. CLL

      * At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy.
      * Less than 1 year between last chemotherapy and progression (i.e. most recent progression free interval <1 year).
      * Not eligible or appropriate for conventional allogeneic SCT
      * Disease responding or stable after most recent therapy (chemotherapy, MoAb)
   4. Mantle cell lymphoma

      * Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT
      * Disease responding or stable after most recent therapy (chemotherapy, MoAb)
      * Relapsed after prior autologous SCT
   5. B-cell prolymphocytic leukemia (PLL) with relapsed or residual disease after at least 1 prior therapy and not eligible for allogeneic SCT.
   6. Diffuse large cell lymphoma or other high-grade NHL, previously identified as CD19+

      * Residual disease after primary therapy and not eligible for autologous SCT
      * Relapsed after prior autologous SCT
      * Beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT
2. Age 1 to 24 years. Patients ages 22-24 will only be enrolled if they are currently being treated at CHOP or another pediatric facility/oncologist
3. Expected survival > 12 weeks
4. Creatinine < 2.5 mg/dl and less than 2.5x normal for age
5. ALT ≤ 5x normal
6. Bilirubin <2.0 mg/dl
7. Any relapse after prior SCT will make patient eligible regardless of other prior therapy
8. Patients with relapsed disease after prior allogeneic SCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and

   1. Have no active GVHD and require no immunosuppression
   2. Are more than 4 months from transplant
9. For those patients who require leukapheresis for T cell collection (i.e. no previously collected product exists), adequate venous access for apheresis or eligible for appropriate catheter placement, and no other contraindications for leukapheresis
10. Voluntary informed consent is given
11. Patients with CNS3 disease will be eligible if CNS disease is responsive to therapy (at infusion)

Exclusion Criteria:

1. Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
2. Uncontrolled active infection
3. Active hepatitis B or hepatitis C infection
4. Concurrent use of systemic steroids at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of inhaled steroids, or hydrocortisone for physiological replacement in patients with adrenal insufficiency are permitted as well
5. Presence of grade 2-4 acute or extensive chronic GVHD
6. Under treatment for GVHD
7. Previous treatment with any gene therapy products
8. Any uncontrolled active medical disorder that would preclude participation as outlined.
9. HIV infection.
10. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2011-08-17 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Grupp, MD,PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- CHOP - http://www.chop.edu/service/oncology/pediatric-cancer-research/cart-19-trial.html, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gofshteyn JS, Shaw PA, Teachey DT, Grupp SA, Maude S, Banwell B, Chen F, Lacey SF, Melenhorst JJ, Edmonson MJ, Panzer J, Barrett DM, McGuire JL. Neurotoxicity after CTL019 in a pediatric and young adult cohort. Ann Neurol. 2018 Oct;84(4):537-546. doi: 10.1002/ana.25315. Epub 2018 Sep 26. PMID 30178481
- [Derived] Fitzgerald JC, Weiss SL, Maude SL, Barrett DM, Lacey SF, Melenhorst JJ, Shaw P, Berg RA, June CH, Porter DL, Frey NV, Grupp SA, Teachey DT. Cytokine Release Syndrome After Chimeric Antigen Receptor T Cell Therapy for Acute Lymphoblastic Leukemia. Crit Care Med. 2017 Feb;45(2):e124-e131. doi: 10.1097/CCM.0000000000002053. PMID 27632680
- [Derived] Maude SL, Frey N, Shaw PA, Aplenc R, Barrett DM, Bunin NJ, Chew A, Gonzalez VE, Zheng Z, Lacey SF, Mahnke YD, Melenhorst JJ, Rheingold SR, Shen A, Teachey DT, Levine BL, June CH, Porter DL, Grupp SA. Chimeric antigen receptor T cells for sustained remissions in leukemia. N Engl J Med. 2014 Oct 16;371(16):1507-17. doi: 10.1056/NEJMoa1407222. PMID 25317870

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CART-19 T Cells
Started | 73 (Number of enrolled subjects)
Intervention | 62
Completed | 21 (Follow up phase completed as per protocol)
Not Completed | 52
Not completed — Adverse Event | 3
Not completed — Disease progression | 27
Not completed — Withdrawal by Subject | 1
Not completed — Administrative problem | 1
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — New cancer therapy | 16
Not completed — Manufacturing failure | 1

BASELINE CHARACTERISTICS:
Population: Subjects that received study treatment
Arm/Group | CART-19 T Cells
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 53
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Study Related Adverse Events.
Description: Inclusive of any events that are "possibly", "likely", or "definitely" related to study treatment any time from the first day of study treatment until week 24.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CART-19 T Cells
Number analyzed (Participants) | 62
Participants | 59

2. Secondary Outcome: The Number of Subjects With a Successful Product Manufactured
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CART-19 T Cells
Number analyzed (Participants) | 62
Participants | 60

3. Secondary Outcome: Number of Subjects With Complete Remission (CR).
Description: Complete remission rate for subjects with Non-CNS3 ALL.
  National Comprehensive Cancer Network standard response criteria, which define complete remission (CR) as ,5% bone marrow blasts by morphologic determination, with no evidence of extramedullary disease or refractory disease.
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CART-19 T Cells
Number analyzed (Participants) | 62
Participants | 16

4. Secondary Outcome: Number of Subjects With Complete Remission With Incomplete Blood Count Recovery (CRi).
Description: as for outcome 3
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CART-19 T Cells
Number analyzed (Participants) | 62
Participants | 38

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | CART-19 T Cells
All-Cause Mortality (participants affected / at risk) | 2/73
Serious Adverse Events (participants affected / at risk) | 58/73
Other Adverse Events (participants affected / at risk) | 62/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CART-19 T Cells (N=73)
Febrile neutropenia (Blood and lymphatic system disorders) | 46
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 6
Coagulopathy (Blood and lymphatic system disorders) | 3
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 4
Bradycardia (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 15
Vascular stent thrombosis (General disorders) | 1
Cytokine release syndrome (Immune system disorders) | 52
Anaphylactic reaction (Immune system disorders) | 1
Device related infection (Infections and infestations) | 5
Lung infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Varicella zoster virus infection (Infections and infestations) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 17
Seizure (Nervous system disorders) | 4
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Speech disorder (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 24
Capillary leak syndrome (Vascular disorders) | 10
Haemolysis (Blood and lymphatic system disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Facial pain (General disorders) | 1
Pain (General disorders) | 3
Bk virus infection (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Stomatococcal infection (Infections and infestations) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Unresponsive to stimuli (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Pyomyositis (Infections and infestations) | 1
Staphylococcal skin infection (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Complication associated with device (General disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Central nervous system haemorrhage (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CART-19 T Cells (N=73)
Febrile neutropenia (Blood and lymphatic system disorders) | 10
Lymphopenia (Blood and lymphatic system disorders) | 50
Splenomegaly (Blood and lymphatic system disorders) | 5
Sinus tachycardia (Cardiac disorders) | 12
Tachycardia (Cardiac disorders) | 30
Conjunctival haemorrhage (Eye disorders) | 4
Diplopia (Eye disorders) | 4
Photophobia (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 21
Constipation (Gastrointestinal disorders) | 10
Diarrhoea (Gastrointestinal disorders) | 35
Haematochezia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 45
Vomiting (Gastrointestinal disorders) | 48
Chills (General disorders) | 27
Fatigue (General disorders) | 29
Pain (General disorders) | 28
Pyrexia (General disorders) | 15
Hepatomegaly (Hepatobiliary disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 13
Cytokine release syndrome (Immune system disorders) | 5
Hypogammaglobulinaemia (Immune system disorders) | 42
Otitis media (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 4
Respiratory syncytial virus infection (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 11
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 11
Activated partial thromboplastin time prolonged (Investigations) | 22
Alanine aminotransferase increased (Investigations) | 45
Aspartate aminotransferase increased (Investigations) | 46
Blood bilirubin increased (Investigations) | 15
Blood creatinine increased (Investigations) | 23
Blood fibrinogen decreased (Investigations) | 11
Blood immunoglobulin A decreased (Investigations) | 5
Blood immunoglobulin M decreased (Investigations) | 5
Blood uric acid increased (Investigations) | 11
Haemoglobin decreased (Investigations) | 57
International normalised ratio increased (Investigations) | 16
Lipase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 6
Neutrophil count decreased (Investigations) | 56
Platelet count decreased (Investigations) | 54
Weight decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 58
Decreased appetite (Metabolism and nutrition disorders) | 43
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hyperphosphataemia (Metabolism and nutrition disorders) | 22
Hyperuricaemia (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 11
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 15
Metabolic acidosis (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Pain in jaw (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 46
Tremor (Nervous system disorders) | 4
Device occlusion (Product Issues) | 4
Anxiety (Psychiatric disorders) | 5
Confusional state (Psychiatric disorders) | 15
Insomnia (Psychiatric disorders) | 8
Haematuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Reproductive system and breast disorders) | 16
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 10
Dermatitis (Skin and subcutaneous tissue disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 9
Pruritus generalised (Skin and subcutaneous tissue disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 6
Rash papular (Skin and subcutaneous tissue disorders) | 8
Skin lesion (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 13
Hypotension (Vascular disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 3
Vision blurred (Eye disorders) | 3
Gingival bleeding (Gastrointestinal disorders) | 3
Mouth haemorrhage (Gastrointestinal disorders) | 3
Catheter site haemorrhage (General disorders) | 3
Catheter site pain (General disorders) | 3
Complication associated with device (General disorders) | 3
Face oedema (General disorders) | 3
Generalised oedema (General disorders) | 3
Withdrawal syndrome (General disorders) | 3
Seasonal allergy (Immune system disorders) | 3
Clostridium difficile colitis (Infections and infestations) | 3
Escherichia urinary tract infection (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Transfusion reaction (Injury, poisoning and procedural complications) | 3
Amylase increased (Investigations) | 3
Prothrombin time prolonged (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Depression (Psychiatric disorders) | 3
Irritability (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT01626495/Prot_SAP_000.pdf